CLINICAL TRIAL: NCT01681745
Title: Probe Configuration and Time-Temperature Dose Ranging for Understanding of Skin Lesion Effects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MYO-0535
Record Dates: First submitted 2012-09-05; First posted 2012-09-10 (Estimated); Results first posted 2021-03-11 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Histological Response of Tissue to Cold

STUDY DESIGN:
Intervention Model Description: Subjects' abdomens treated with Myoscience device (cryoneurolysis) at various timepoints prior to an abdominoplasty. Skin examined visually and resected for histological examination.
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cryo-Touch Treatment (Experimental): Initial treatment with Cryo-Touch III and three optional re-treatments (up to 4 treatments) performed 68 days to 1 day prior to abdominoplasty.
  Interventions: Device: Cryo-Touch III

INTERVENTIONS:
Device: Cryo-Touch III
  Other Names: PCP 1.0

SUMMARY:
This study is designed to characterize the biological response of the epidermis, dermis and subcutaneous tissue to treatment with the Myoscience Cryo-Touch III system.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 to 70 years old
* Subject is willing and able to give written informed consent.
* Subject is committed to undergo an abdominoplasty procedure independent of this study.
* Subject is willing and able to comply with study instructions and commit to all visits for the duration of the study.
* Subject is in good general health and free of any disease state or physical condition that might impair evaluation or which in the investigator's opinion, expose the subject to an unacceptable risk by study participation.

Exclusion Criteria:

* Subject is currently enrolled in an investigational drug or a device study that specifically targets the abdominal area.
* Subject currently smokes.
* Subject has a clotting disorder and/or has used an anticoagulant (e.g., warfarin, clopidogrel, etc.) within seven (7) days prior to administration of the device.
* Subject has used oral or inhaled steroids in the last 14 days and/or has been a chronic user of inhaled or oral steroids in the past such that the investigator feels subject may have compromised wound healing.
* Subject has used topical steroids in the abdominal area within the last 30 days.
* Subject is on any systemic immunosuppressive therapy.
* Subject has had prior surgery and/or treatment that alters the subcutaneous anatomy of the target treatment sites: liposuction, cryolipolysis, or high-intensity focused ultrasound.
* History of abdominal hernia.
* Subject has any of the following conditions:
* Allergy or intolerance to lidocaine,
* Other local skin condition (e.g., skin infection) at target treatment site,
* Any physical or psychiatric condition that in the investigator's opinion would prevent adequate study participation.
* Chronic medical condition or use of medication that in the investigator's opinion would affect study participation or wound healing (such as diabetes, hepatitis, HIV, etc.).
* Subject is known to be noncompliant or is unlikely to comply with the requirements of the study protocol (e.g., due to alcoholism, drug dependency, mental incapacity) in the opinion of the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-06-01 (Actual); Primary Completion 2015-04-01 (Actual); Study Completion 2015-04-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- 77 Plastic Surgery, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During transfer and acquisition of study record by sponsors, no study data has been located and all efforts to locate study data have been exhausted. Therefore, no study data is available to report at this time.
Period: Overall Study
Arm/Group | Cryo-Touch Treatment
Started | 0
Completed | 0
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: During transfer and acquisition of study record by sponsors, no study data has been located and all efforts to locate study data have been exhausted. Therefore, no study data is available to report at this time.
Arm/Group | Cryo-Touch Treatment
Number analyzed (Participants) | 0
Age, Continuous [unit: years]
Sex: Female, Male

OUTCOME MEASURES:

1. Primary Outcome: Biological Tissue Response
Description: The biological response of the treated tissue by the Cryo-Touch III or Cryo-Touch IV device was determined through gross pathology and histological assessment.
Time Frame: 7 days
Population: as for baseline characteristics
Arm/Group | Cryo-Touch Treatment
Number analyzed (Participants) | 0

2. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs) and Unanticipated Adverse Events (UADEs)
Description: All anticipated observations, adverse events and SAEs/UADEs were assessed. Incidence of serious adverse events (SAEs) and unanticipated adverse device effects (UADEs) were recorded.
Time Frame: 7 days
Population: as for baseline characteristics
Arm/Group | Cryo-Touch Treatment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: During transfer and acquisition of study record by sponsors, no study data has been located and all efforts to locate study data have been exhausted. Therefore, no study data is available to report at this time.
Arm/Group | Cryo-Touch Treatment
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
During transfer and acquisition of study record by sponsors, no study data has been located and all efforts to locate study data have been exhausted. Therefore, no study data is available to report at this time.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No